CLINICAL TRIAL: NCT06504563
Title: Relationship Between Kinesthetic Perception, Motor Competence, Physical Fitness and Emotional Intelligence in Obese School Children
Brief Title: Relationship Between Kinesthetic Perception, Motor Competence, Physical Fitness and Emotional Intelligence in Children
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0781
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Children
Keywords: Kinesthetic perception,; motor competence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The benefits of an active lifestyle and physical fitness extend to physical, mental, and social aspects of well-being, including improved cardiopulmonary health, concentration, and self-confidence. The World Health Organization recommends 60 minutes of daily activity to combat childhood obesity, which is influenced by factors like lack of exercise, poor diet, and sedentary behaviors. Obesity negatively impacts children's kinesthetic perception, motor skills, and emotional resilience, crucial for their nervous system development. This study aims to explore the relationship between these factors in obese school-age children.

DETAILED DESCRIPTION:
The data will be collected by both subjective and objective assessments. The data collection will be organized at the premises of the participating schools during the time allocated for physical education and breaks. Consent will be taken from each participant before any assessment. The data will be collected included anthroprometric and demographics included sex, age, class/grade level, height, weight, BMI (calculated as the weight divided by the square of height). Measurement tools such as, PMSC will be used to assess motor competence and physical fitness in young children. It is a performance based tool, PMSC will assess children's fundamental locomotion skills such as catching, running, kicking, jumping forward, skipping and hitting ball with one hand. Each question will be scored as 'good' or 'not as good'. Kinesthetic perception will be assessed by Nelson hand reaction time. It is a performance based activity. It will test the subject's kinesthetic perception visually, auditory senses and tactile senses. Emotional Intelligence will be assessed using PANAS tool.

ELIGIBILITY:
Inclusion Criteria:

* Age of the participants 10 to 15 years
* Male and female will be included.
* Obese Class 1, class 2, class 3

Exclusion Criteria:

* Children who have high risk level and poor safety as it pertains to physical activity.
* Children with disabilities that are limited in their ability to understand the testing instructions or the performance of the activities (e.g., cognitive impairments, gross motor impairments etc.). •. Children with any kind of disability and congenital deformity

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Obese children are recruited, male and female. The age limit is from 10 years to 15 years
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Kinesthetic Perception | 8 weeks
  Kinesthetic perception will be assessed by Nelson hand reaction. The term Reaction time is the interval of time between the presentation of the stimulus and the initiation of response. Motor competence will be assessed using the pictorial scale of Perceived Movement Skill Competence (PMSC) for young children. Emotional intelligence will be assessed by using PANAS tool. Affect indicates people's positive and negative emotions and is composed of Positive Affect (PA) or pleasant emotions and Negative Affect (NA) or unpleasant emotions.
Physical fitness | 8 weeks
  endurance will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Bakhtiar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jebeile H, Kelly AS, O'Malley G, Baur LA. Obesity in children and adolescents: epidemiology, causes, assessment, and management. Lancet Diabetes Endocrinol. 2022 May;10(5):351-365. doi: 10.1016/S2213-8587(22)00047-X. Epub 2022 Mar 3. PMID 35248172